CLINICAL TRIAL: NCT00906841
Title: Phase II Study of Evaluation of Fractionated Radio-immunotherapy With 90Y-DOTA-hLL2 as a Consolidation Therapy After First Line of Chemotherapy in Patients Older Than 60 With Disseminated Diffuse Large B-cell Lymphoma
Brief Title: Study of 90Y-DOTA-hLL2 as a Consolidation Therapy After R-CHOP in Patients With Diffuse Large B-cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: completed recruitment of patients on 15 december 2010
Sponsor: French Innovative Leukemia Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIT90Y-DOTA-hLL2
Record Dates: First submitted 2009-05-18; First posted 2009-05-21 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: B-cell Lymphoma
Keywords: Disseminated diffuse large B-cell lymphoma; first line treatment; R CHOP; 90Y-DOTA-hLL2; Patients older than 60 years
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Consolidation Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 90Y-DOTA-hLL2 (Experimental): Fractionated RIT (8 weeks after the end of R-CHOP: 2 injections of 15 mCi/m2 of 90Y-DOTA-hLL2 and hLL2 at day 1 and day 8)
  Interventions: Drug: 90Y-DOTA-hLL2

INTERVENTIONS:
Drug: 90Y-DOTA-hLL2 — Consolidation : Fractionated RIT (8 weeks after the end of R-CHOP: 2 injections of 15 mCi/m2 of 90Y-DOTA-hLL2 and hLL2 at day 1 and day 8)
  Other Names: consolidation

SUMMARY:
Phase II, multi-centric, open-label, study.

Disseminated diffuse large B-cell lymphoma in patients older than 60: evaluation of fractionated radio-immunotherapy with 90Y-DOTA-hLL2 as a consolidation therapy after first line of chemotherapy.

DETAILED DESCRIPTION:
Initial treatment: 6 courses of CHOP-R 14 with evaluation of response before C4 (observation of no change or progression at this time will get the patient off study).

Consolidation : fractionated RIT (8 weeks after the end of R-CHOP: 2 injections of 15 mCi/m2 of 90Y-DOTA-hLL2 and hLL2 at day 1 and day 8).

ELIGIBILITY:
Inclusion Criteria:

* Age > 60 and < 80 years
* Non eligible for stem cell transplantation
* CD20 diffuse large B-cell lymphoma according to the WHO classification
* Bulky stage I and II > ou =7 cm and stage III and IV
* Performance status 0 - 2
* Creatinine clearance >ou = 50 ml/min (Cockroft formula).
* Serum bilirubin < ou =30 mmol/l
* Leucocytes > ou =3 G/l, granulocytes > ou = 1,5 G/l, platelets >ou= 100 G/L.
* HIV negative
* Written informed consent

Exclusion Criteria:

* Age < 60 years and > 80 years
* Other types of lymphomas except CD20+ diffuse large B-cell lymphoma according to the WHO classification
* Histologic transformation of low grade lymphoma (Involvement of the bone marrow by small B-cell lymphoma will not lead to exclusion of the patient)
* Primary lymphoma of the central nervous system and transformed gastro intestinal MALT lymphoma
* Meningeal involvement
* Bone marrow involvement > 25% after R-CHOP
* Aggressive post-transplantation lymphoma
* Absence of CD20 expression on tumor cells
* Non bulky stages I et II
* HIV positive
* Active Hepatitis B or C
* Left ventricular ejection fraction < 50%.
* Contra-indication to R-CHOP treatment
* Previous or concurrent second malignancy except for adequately treated basal cell carcinoma of the skin, curatively treated in situ carcinoma of the cervix, curatively treated solid cancer, with no evidence of disease for at least 5 years
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Participation at the same time in another study in which investigational drugs are used
* Absence of written informed consent

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-10; Primary Completion 2016-03 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Event free survival (EFS) | EFS post treatment (at 2 years)

SECONDARY OUTCOMES:
Objective disease response (CR, CRu and PR), SD and disease progression | OS after treatment
Duration of response | Time interval from the date on which a response (CR, CRu and PR)
Time to disease progression | Time interval from the date from initial of study treatment until the date on which disease progression is documented

CONTACTS AND LOCATIONS:
Overall Officials: Françoise KRAEBER BODERE, MDPD, Principal Investigator — French Innovative Leukemia Organisation; Pierre SOUBEYRAN, MD, Principal Investigator — French Innovative Leukemia Organisation
Locations (1):
- Chu/Clcc Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kraeber-Bodere F, Pallardy A, Maisonneuve H, Campion L, Moreau A, Soubeyran I, Le Gouill S, Tournilhac O, Daguindau E, Jardel H, Morineau N, Bouabdallah K, Gyan E, Moles MP, Gressin R, Berthou C, Sadot S, Moreau P, Deau B, Bodet-Milin C, Cazeau AL, Garin E, Salaun PY, Vuillez JP, Gouilleux-Gruart V, Barbet J, Wegener WA, Goldenberg DM, Lamy T, Soubeyran P. Consolidation anti-CD22 fractionated radioimmunotherapy with 90Y-epratuzumab tetraxetan following R-CHOP in elderly patients with diffuse large B-cell lymphoma: a prospective, single group, phase 2 trial. Lancet Haematol. 2017 Jan;4(1):e35-e45. doi: 10.1016/S2352-3026(16)30168-5. Epub 2016 Dec 8. PMID 27964867
- See also: FILO Internet site — http://www.filo-leucemie.org